CLINICAL TRIAL: NCT02062970
Title: Interest of the Balance of Pro-coagulating and Profibrinolytis Activities of the Microparticles (MP) in the Prognosis of Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A01251-44; 2013-36 (Other: Assistance Publique des Hôpitaux de Marseille)
Record Dates: First submitted 2013-11-28; First posted 2014-02-14 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: the Coagulolytic Balance; the Mortality Rate; the Performance Used to Evaluate the Principal Objective Are Technical Performances, Sensibility and Specificity of the Tests
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- septic shock patients suffering (Experimental): blood sample done in a population whom suffer of septic shock
  Interventions: Biological: blood draw

INTERVENTIONS:
Biological: blood draw

SUMMARY:
Septic shock is a clinical syndrome occurring in 10 to 20% of patients admitted in ICV. Mortality associated to septic shock varies from 30 to 50%. It follows a systemic response of the organism to a severe infection, associated with a circulatory failure marker by an arterial hypotension and a vascular hyperactivity to vasoconstrictor agents.

The mechanisms involved on one hand an activation of white blood cells inflammatory system and the vascular inflammatory system; and on the other hand on imbalance in hemostatis characterized by an activation of the coagulation and an inappropriate fibrinolysis leading to a disruption of microcirculation in the context of a disseminated intravascular coagulation (DIVC).

This inflammatory and thrombotic cellular activation is strongly associated with the phenomenon of vesiculation; leading to the production of cellular microparticles (MP) by blood cells and vascular cells.

MP are membranous vesicles, resulting in the reassortment of membrane phospholides in response to an activation of cellular apoptosis. They have been initially described as new actors of hemostatis. Indeed, the expression of phospholipid serine and tissular factor (TF) confer them a procoagulating activity, which increases in patients undergoing septic shock.

The finding of a fibriniolytic activity of the cellular MP suggests the existence of compensating mechanisms with a procoagulating activity. This confers to MP a key-role in the control of the coagulolytic balance.

Our recent researches suggest that endothelial and white blood cells MP produce in vivo plasmin.

They carry into the main circulation a fibrinolytic activity which is partially beyond the physiological inhibitors activity (PAI-1, x 2 antiplasmin). Preliminary findings show that this ability of plasmin generation is important in patients affected with septic shock.

Our hypothesis is that an increase in plasmin generation by MP compensates the risk of occurrence of microthrombosis, modulating therefore the vital prognosis of patients with septic shock.

The coagulolytic balance of MP, which is resulting of their own procoagulating and fibrinolytic activities could claim the status of new pronostic marker relevant in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patient with septic shock

Exclusion Criteria:

* age under 18 yo
* pregnant woman
* septic shock since more than 24 hours
* patient hospitalized for cardiac arrest
* immunocompromised patients
* patient in whom the stop of active therapeutic is discuss
* patient treated with an anti-coagulant at therapeutic dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the interest of the measure of the coagulolytic balance, dependant of the circulating MP in the prognostic of mortality in a population of subjects presenting a septic shock. | 36 month
  The outcome of the study is to evaluate the interest of the measure of the coagulolytic balance, dependant of the circulating MP in the prognostic of mortality in a population of subjects presenting a septic shock. The objective is to evaluate the performance of this dosage while estimating the ROC-surve.
  In this present project:
  • the coagulolytic balance dependant of the MP is defined by the ratio between the activity of production of thrombin of circulating MP expressed by a speed in nM thrombin per minutes : and the activity of production of plasmin of circulating MP expressed by a speed in DD per minutes measured at inclusion of the subjects ; within 48 hours after diagnosis ;

CONTACTS AND LOCATIONS:
Overall Officials: Mondoloni Loic, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique des Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Lacroix R, Judicone C, Souab KH, Bonifay A, Loundou A, Bouriche T, Cointe S, Vallier L, Abdili E, Arnaud L, Robert S, Poncelet P, Grosdidier C, Morange P, Cochery-Nouvellon E, Bouvier S, Gris JC, Lefrant JY, Leone M, Albanese J, Dignat-George F. The Procoagulant and Fibrinolytic Balance of Extracellular Vesicles Predicts Mortality in Septic Shock Patients. J Extracell Vesicles. 2025 Jun;14(6):e70073. doi: 10.1002/jev2.70073. PMID 40560804